CLINICAL TRIAL: NCT05381415
Title: Effect on Bronchodilatation Response and Ventilation Heterogeneity of Different Inhalation Volumes in COPD: the BREATH COPD Study
Brief Title: Effect on Bronchodilation Response and Ventilation Heterogeneity of Different Inhalation Volumes in COPD
Acronym: BREATH COPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Collaborators: Department of Clinical and Surgical Pathophysiology and Transplantation, University of Milan (Unknown)
Responsible Party: Principal Investigator, Pierachille Santus, MD, PhD, Professor of Pulmonary Medicine, University of Milan
Other Study IDs: BREATHCOPD2022
Record Dates: First submitted 2022-05-04; First posted 2022-05-19 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: COPD; Lung Injury
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with COPD: Patients with COPD diagnosis (VEMS/FVC after bronchodilatation <0.7) will be enrolled in a stable state of disease, diagnosed from at least 12 months [GOLD].
  Each patient will be studied during three visits. In the first visit it will be established the patient eligibility. Furthermore, the patient will be able to familiarize with the experimental procedure. Chronic inhalation therapy will be suspended 24 (long action) and 8 (short action) hours before the second and third visit. If a patient is on tiotropium bromide, it will be required to be suspended 7 days before the visit.
  During the second and third visit, which will be scheduled 30 days one from another, the patient will be asked to inhale the bronchodilator (salbutamol pMDI, 400 µg) with a spacer from VR or FRC, in a random order. Before and after the administration it will be asked to the patient to execute a spirometry, a plethysmography, a lung diffusion test, and the NEP technique.
  Interventions: Other: Inhalation of bronchodilation therapy at FRC; Other: Inhalation of bronchodilation therapy at RV

INTERVENTIONS:
Other: Inhalation of bronchodilation therapy at FRC — the patient will be asked to inhale the bronchodilator (salbutamol pMDI, 400 µg) with a spacer from FRC (functional residual capacity, in a random order, with the assistance of an operator. The spacer will be connected to a Fleish flowmeter placed in series with the pMDI device.
  The valve included in the spacer will guarantee that only the air inhaled by the patient will pass through the flowmeter, reducing the risk of contamination. In both cases a low inspiratory flux and a period of apnea after inhalation of 10 seconds will be used. Before and after the administration it will be asked to the patient to execute a spirometry, a plethysmography, a lung diffusion test, and the NEP technique. These will allow the characterization of the bronchodilator effect in terms of static and dynamic volumes, heterogeneity of ventilation distribution and volume of closure, expiration flux-limitation.
Other: Inhalation of bronchodilation therapy at RV — the patient will be asked to inhale the bronchodilator (salbutamol pMDI, 400 µg) with a spacer from VR , with the assistance of an operator. The spacer will be connected to a Fleish flowmeter placed in series with the pMDI device.
  The valve included in the spacer will guarantee that only the air inhaled by the patient will pass through the flowmeter, reducing the risk of contamination. In both cases a low inspiratory flux and a period of apnea after inhalation of 10 seconds will be used. Before and after the administration it will be asked to the patient to execute a spirometry, a plethysmography, a lung diffusion test, and the NEP technique. These will allow the characterization of the bronchodilator effect in terms of static and dynamic volumes, heterogeneity of ventilation distribution and volume of closure, expiration flux-limitation.

SUMMARY:
During bronchodilator tests, it's common to ask patients with asthma or chronic obstructive pulmonary disease (COPD) to take bronchodilator therapy by inhaling after a maximal exhalation, when the respiratory system volume equals the residual volume. The same maneuver is required for the chronic therapy.

Nevertheless, in patients with COPD the distribution of ventilation is more heterogeneous, especially when lung volumes are closer to residual volume . It is therefore predictable that the distribution of air volume containing bronchodilator that has been inhaled at residual volume is more heterogeneous than at higher volumes, such as at functional residual capacity. Accordingly, the bronchodilator can be preferentially distributed in more open airways than in less patent ones, with a heterogeneous distribution of the medication. Therefore, the overall bronchodilation should be greater when the drug inhalation is performed at functional residual capacity than at residual volume.

It is common knowledge that the effectiveness of bronchodilator therapy with pMDI in subjects with COPD is greatly affected by the inhalation technique, which can be difficult to perform for many patients. Therefore, in addition to the possibility that inhalation of bronchilation therapy at residual volume could lower the drug effectiveness, this maneuver complicates the sequence of actions required to the patient, enhancing the risk of errors and decreasing the aderence to treatment.

The aim of this study is to investigate whether the inhalation of a bronchodilator at different lung volumes can affect its effectiveness in terms of respiratory function, in patients with COPD.

Assuming that the bronchodilator effectiveness is equal or greater when inhaled at functional residual capacity rather than at residual volume, the inhalation maneuver can be simplified for patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* age above 40 years old;
* history of smoking equal or above 10 PKYs;
* VEMS after bronchodilatation ≤ 70%,
* medical Necessity to perform a bronchodilatation test.

Exclusion Criteria:

* history of bronchial asthma or other chronic respiratory diseases such as pulmonary fibrosis;
* uncontrolled cardiovascular diseases at the time of the visit;
* current pregnancy;
* incapacity to execute lung function tests for cognitive impairment, substance abuse or claustrophobia;
* known hypersensitivity or intolerance to salbutamol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD diagnosis (VEMS/FVC after bronchodilatation <0.7) will be enrolled in a stable state of disease, diagnosed from at least 12 months [GOLD].
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of bronchodilation therapy inhaled at Functional Residual Capacity (FRC) on Forced Expiratory Volume in 1 second (FEV1) | 1 year
  Assuming that the bronchodilator effectiveness is equal or greater when inhaled at functional residual capacity rather than at residual volume, the inhalation maneuver can be simplified for patients with COPD.

SECONDARY OUTCOMES:
Effects on change in phase III slope of the closing volume curve | 1 year
  Efficacy of bronchodilation therapy inhaled at FRC on reducing phase III slope of the closing volume, as compared to bronchodilation therapy inhaled at RV
Effects on forced vital capacity (FVC) | 1 year
  Efficacy of bronchodilation therapy inhaled at FRC on static and dynamic lung volumes as compared to bronchodilation therapy inhaled at RV
Effects on vital capacity (VC) | 1 year
  Efficacy of bronchodilation therapy inhaled at FRC on static and dynamic lung volumes as compared to bronchodilation therapy inhaled at RV
Effects on residual volume (RV) | 1 year
  Efficacy of bronchodilation therapy inhaled at FRC on static and dynamic lung volumes as compared to bronchodilation therapy inhaled at RV
Effects on total lung capacity (TLC) | 1 year
  Efficacy of bronchodilation therapy inhaled at FRC on static and dynamic lung volumes as compared to bronchodilation therapy inhaled at RV
Effects on sensation of dyspnea as measured by modified Medical Research Council (mMRC) score | 1 year
  Efficacy of bronchodilation therapy at functional residual capacity on sensation of dyspnea
Effects on specific airway resistance (sRAW) | 1 year
  Efficacy of bronchodilation therapy at functional residual capacity on specific pulmonary resistances

CONTACTS AND LOCATIONS:
Locations (1):
- L. Sacco Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No